CLINICAL TRIAL: NCT06038045
Title: PROSPER- Electronic Patient Reported OutcomeS to Empower Patients rEcoveR
Brief Title: Measuring the Recovery of Barts Health Patients With Electronic Follow-up
Acronym: PROSPER
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 318066
Record Dates: First submitted 2023-08-31; First posted 2023-09-14 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Surgery; Critical Illness; Trauma
MeSH Terms: conditions — Critical Illness; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
More and more people are surviving emergency, life-threatening illnesses. However, survival often comes at a cost to patients' wellbeing. Many suffer from being so ill in ways not necessarily related to their original illness. Patients struggle with their normal activities of daily living or to do the job they did before. They struggle to live independently, to enjoy a normal diet, or to be pain-free. This leads to a decrease in their quality of life, placing a burden on families. Investigators don't have a good method of highlighting and representing the issues faced by these patients. Investigators have recently implemented a service innovation project, using an an app-based questionnaire in two groups (patients that survive emergency surgery, and those who survive critical illness) to highlight these problems early, so that individuals are offered the right help and services to return to living their lives as fully as possible. Patients will be asked to fill in an electronic (on-line) questionnaire while in hospital, and at 1 and 6 months afterwards.

Along side this investigators intend to perform a qualitative assessment of the value and acceptability of this project. Investigators will interview patients approximately 2-3 weeks after the questionnaire completion at 1 and 6 months to determine how easy it was to use, how acceptable the process was and how well it described and highlighted their problems.

If this system works, it would become part of routine care, extended to patients admitted as emergencies to hospital, and used to develop a national program for all UK hospital patients

DETAILED DESCRIPTION:
This is a qualitative study, with data collected through semi-structured interviews with patients and clinical staff with experience of using the ePRO system. Topic guides for both patients and clinicians have been developed based upon previous similar studies and with input from our study PPI group.

The patients for qualitative study will be consented by the coordinator. This will be done when the patients are invited to participate in the PROSPER study. The ePRO project is a service evaluation project registered with the Clinical Effectiveness Unit (CEU). The sample for qualitative study will be based on age, gender, ethnicity, language spoken, digital literacy and reason for admission. Patients who consent to participate will be interviewed twice about their experience of using the ePRO system. Interviews will be done approximately 2-3 weeks after the ePRO questionnaire completion time points of 1 and 6 months respectively. Interviews will follow the interview topic guide, with semi-structured questions exploring both the research objectives as above, will be conducted on the telephone and will be audio recorded and transcribed. Clinicians and health care staff will also be interviewed to assess their perception of usefulness of the electronic questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing emergency laparotomy, regardless of admission to the Adult Critical Care Unit.
* Patients requiring Level 3 care admitted to the Adult Critical Care Unit with length of stay of >56 hours
* Clinical staff involved in the pathway of care affected by the ePRO.
* Purposive sampling to include patients based on age, gender, ethnicity, language spoken, digital literacy and reason for admission

Exclusion Criteria:

Those patients <18 years of age

* Those not expected to survive 3 months post discharge; as per clinical decision making
* Patients unable to consent to and without carers able to consent;

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients that are admitted to the critical care wards with any indication, and those above the age of 18 years and able to consent for the study.
  The PI will adopt a purposive sampling method to ensure that age, gender and ethnicity is equally represented in the population.
  Furthermore, the health care staff including clinicians, and follow- up clinic staff, physiotherapists, dieticians/nutritionist alike and staff involved in healthcare will be interviewed for their feedback on the questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
This is a qualitative study exploring the feasibility and acceptability of the electronic HRQoL | 6 months to one year
  Purposive sampling will be carried out on the patient population those filling in online questionnaires and health care staff involved in patient care. Their views will be recorded to assess the suitability and acceptability of the digital questionnaires. The outcome will be responses to the semi structured interview. These data will be analysed to derive themes, using the saturation method.
  Since August 2024, we have introduced an online questionnaire based on the feedback of a few patients.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Der Wees PJ, Nijhuis-Van Der Sanden MW, Ayanian JZ, Black N, Westert GP, Schneider EC. Integrating the use of patient-reported outcomes for both clinical practice and performance measurement: views of experts from 3 countries. Milbank Q. 2014 Dec;92(4):754-75. doi: 10.1111/1468-0009.12091. PMID 25492603
- [Background] Puthucheary Z, Brown C, Corner E, Wallace S, Highfield J, Bear D, Rehill N, Montgomery H, Aitken L, Turner-Stokes L. The Post-ICU presentation screen (PICUPS) and rehabilitation prescription (RP) for intensive care survivors part II: Clinical engagement and future directions for the national Post-Intensive care Rehabilitation Collaborative. J Intensive Care Soc. 2022 Aug;23(3):264-272. doi: 10.1177/1751143720988708. Epub 2021 Feb 1. PMID 36033242
- [Background] Major ME, van Nes F, Ramaekers S, Engelbert RHH, van der Schaaf M. Survivors of Critical Illness and Their Relatives. A Qualitative Study on Hospital Discharge Experience. Ann Am Thorac Soc. 2019 Nov;16(11):1405-1413. doi: 10.1513/AnnalsATS.201902-156OC. PMID 31394924
- [Background] Law J, Welch C, Javanmard-Emamghissi H, Clark M, Bisset CN, O'Neil P, Moug SJ; ELF study group. Decision-making for older patients undergoing emergency laparotomy: defining patient and clinician values and priorities. Colorectal Dis. 2020 Nov;22(11):1694-1703. doi: 10.1111/codi.15165. Epub 2020 Jun 21. PMID 32464712
- [Background] Vilches-Moraga A, Rowley M, Fox J, Khan H, Paracha A, Price A, Pearce L. Emergency laparotomy in the older patient: factors predictive of 12-month mortality-Salford-POPS-GS. An observational study. Aging Clin Exp Res. 2020 Nov;32(11):2367-2373. doi: 10.1007/s40520-020-01578-0. Epub 2020 May 24. PMID 32449105
- [Background] Poulton TE, Moonesinghe R, Raine R, Martin P; National Emergency Laparotomy Audit project team. Socioeconomic deprivation and mortality after emergency laparotomy: an observational epidemiological study. Br J Anaesth. 2020 Jan;124(1):73-83. doi: 10.1016/j.bja.2019.08.022. PMID 31860444
- [Background] Ray S, Laur C, Golubic R. Malnutrition in healthcare institutions: a review of the prevalence of under-nutrition in hospitals and care homes since 1994 in England. Clin Nutr. 2014 Oct;33(5):829-35. doi: 10.1016/j.clnu.2013.10.017. Epub 2013 Nov 1. PMID 24238787
- [Background] McNelly AS, Rawal J, Shrikrishna D, Hopkinson NS, Moxham J, Harridge SD, Hart N, Montgomery HE, Puthucheary ZA. An Exploratory Study of Long-Term Outcome Measures in Critical Illness Survivors: Construct Validity of Physical Activity, Frailty, and Health-Related Quality of Life Measures. Crit Care Med. 2016 Jun;44(6):e362-9. doi: 10.1097/CCM.0000000000001645. PMID 26974547